CLINICAL TRIAL: NCT02753153
Title: Extraction Socket Management Using Connective Tissue Graft Versus Mucograft®: A Randomized Controlled Trial
Brief Title: Extraction Socket Management Using Connective Tissue Graft Versus Mucograft®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Prof. Dr. France LAMBERT, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2010-1
Record Dates: First submitted 2016-04-14; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Tooth Lost
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mucograft®, Geistlich Biomaterials (Experimental): A Mucograft membrane will be used in state of a connective tissue graft. The dimension of the Mucograft® will be previously calculated according to the site dimensions and inserted into buccal pouch and sutured to be stabilized on the buccal aspect. The membrane is then positioned to cover the socket and inserted and sutured in the palatal pouch by the means of vertical interrupted sutures
  Interventions: Procedure: Test surgical protocol; Procedure: Socket preservation
- Soft tissue graft (Active Comparator)
  Interventions: Procedure: Control surgical protocol; Procedure: Socket preservation

INTERVENTIONS:
Procedure: Control surgical protocol — A connective tissue graft will be harvested to the palate or posterior maxilla tuberosity. The dimension of the graft will be previously calculated according to the socket dimensions. The harvesting site will be made with a single edge incision and sutured with 4.0 silk (uninterrupted suture). The connective tissue graft will be reshaped if necessary to be 1-2mm thick and inserted into buccal pouch and sutured with 2 vertical interrupted sutures to be stabilized on the buccal aspect.
  The connective tissue graft is then positioned to caver the socket and inserted and sutured in the palatal pouch also by the means of vertical interrupted sutures (polypropylen 6.0).
  Arms: Soft tissue graft
Procedure: Test surgical protocol — The filling biomaterial (Bio-Oss®, Geistlich), previously humidified with a saline solution containing doxycycline (1mg/ml) and inserted into the socket without heavy compaction.
  Arms: Mucograft®, Geistlich Biomaterials
Procedure: Socket preservation — An atraumatic extraction will be performed in order to preserve the socket bone wall as well as the cervical soft tissues.
  Split- thickness pockets will be performed 5-6 mm deep buccally and 3-4 mm deep palatally preserving interproximal papillae. The filling biomaterial (Bio-Oss®, Geistlich), previously humidified with a saline solution containing doxycycline (1mg/ml) and inserted into the socket without heavy compaction. At this level of the surgery, the randomization envelope will be open and either the control or the test surgical protocol will be applied.

SUMMARY:
This study aims at assessing the hard and soft tissues remodelling of the alveolar crest after extraction socket managements in the aesthetic areas:

* 3D radiographic evaluation (CT scan) was performed post extraction and 3 months after at the time of implant placement. (Outcomes 1: Hard tissues analyses )
* Impressions, models and 3D analyses of the treated area allowed studying external soft tissue remodeling at different time points after extraction. (Outcomes 2: Soft tissues analyses )

ELIGIBILITY:
Inclusion Criteria:

* Patients needing an extraction in the aesthetic area to be replace with an implant (incisive, canine or premolar)
* Good general health (ASA 1, 2)
* Controlled periodontitis
* No age restriction

Exclusion Criteria:

* Extraction socket with buccal bone defect / buccal bone wall dehiscence
* Smokers > 10 cigarettes per day
* Immune system disease
* Bone disease or treatment by medicines interfering with bone metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Bone remodeling of the buccal and palatal walls using radiographic measurements | 1year
  Bone remodeling of the buccal and palatal walls will be measured in cone beam computerized tomography (CBCT) on the day of extraction, at 3 months after implant placement.

SECONDARY OUTCOMES:
Soft tissue contours measurements by 3D image analyses. | 6months
  Models from the different time points are scanned using 3D-Laser-Scanner and Software (Metalor). 3D reconstructions are matched in order to evaluate 3D and 2D volume changes in extraction sites from baseline to implant placement.

OTHER OUTCOMES:
Explants will be analyzed by X-ray computed microtomography | 1year
Explants will be processed for non-decalcified histology using polymethacrylate (PMMA) resin | 1year
Bone formation histomorphometric evaluation using a semiautomatic image analyzer | 1year

IPD SHARING:
Plan to Share IPD: No